CLINICAL TRIAL: NCT07173712
Title: Regimen Transition After Short-Term Intensive Insulin Therapy in Type 2 Diabetes Mellitus Patients With Inadequate Glycemic Control on Oral Hypoglycemic Agents: A Multicenter, Open-Label, Randomized Controlled Study
Brief Title: Regimen Transition After Short-Term Intensive Insulin Therapy in Type 2 Diabetes
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yanbing Li (Other)
Responsible Party: Sponsor-Investigator, Yanbing Li, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2025-182
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin degludec, insulin aspart drug combination; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iGlarLixi group (Active Comparator)
  Interventions: Drug: CSII; Drug: Insulin glargine /lixisenatide Fixed Ratio Combination
- IDegAsp group (Active Comparator)
  Interventions: Drug: CSII; Drug: Insulin Degludec and Insulin Aspart Injection
- iGlar group (Active Comparator)
  Interventions: Drug: Insulin Glargine (HOE901 - U300); Drug: Metformin

INTERVENTIONS:
Drug: CSII — Short term intensive insulin therapy
  Arms: IDegAsp group; iGlarLixi group
Drug: Insulin glargine /lixisenatide Fixed Ratio Combination — Insulin Glargine and Lixisenatide Injection(I) Treatment for 24 weeks
  Arms: iGlarLixi group
Drug: Insulin Degludec and Insulin Aspart Injection — Insulin Degludec and Insulin Aspart Injection Treatment for 24 weeks
  Arms: IDegAsp group
Drug: Insulin Glargine (HOE901 - U300) — Insulin Glargine Treatment for 24 Weeks
  Arms: iGlar group
Drug: Metformin — Metformin Treatment for 24 weeks
  Arms: iGlar group

SUMMARY:
Failure of oral antidiabetic drugs (OADs) is a frequent challenge in patients with type 2 diabetes mellitus (T2DM), and inadequate long-term glycemic control substantially increases the risk of diabetic complications. Short-term intensive insulin therapy (SIIT) is an established approach to mitigate glucotoxicity; however, the optimal strategy to sustain long-term glycemic benefits after SIIT in T2DM patients with OAD failure remains unclear. To address this gap, we designed a randomized controlled trial to evaluate subsequent treatment options, aiming to identify a simple and effective regimen for patients with poor glycemic control who undergo SIIT.

A total of 324 eligible patients will be enrolled. After screening, previous antidiabetic regimens will be discontinued, and patients will be randomly assigned to the SIIT- iGlarLixi group (A), the SIIT-IDegAsp group (B), or the SIIT-iGlar group (C). All patients will be hospitalized for short-term insulin pump therapy, followed by 24 weeks of treatment: group A with insulin glargine/lixisenatide, group B with insulin degludec/aspart, and group C with insulin glargine U300 plus metformin. During the extension follow-up period, patients in all groups may either continue their assigned regimen or return to their original pre-study therapy. A total of 10 clinic visits are scheduled for each patient throughout the study.

Primary endpoint is proportion of patients achieving glycosylated hemoglobin A1C <7% at 24 weeks.Secondary endpoints include proportion of patients achieving glycosylated hemoglobin A1C <6.5% at 24 weeks; differences in weight gain, hypoglycemic events among treatment groups, and differences in proportion of patients continuing the assigned regimen, glycemic control and body weight at the extension follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes mellitus (T2DM) with a disease duration of >1 year and <15 years.
2. On a stable dose of at least one oral antidiabetic drug (OAD) for ≥3 months.
3. HbA1c at screening: >8.0% if on a single OAD; >7.5% if on more than one OAD (centralized laboratory testing, or results from medical centers participating in the National Glycohemoglobin Standardization Program).
4. Age 18-70 years.
5. Body mass index (BMI) 20-35 kg/m².
6. Able and willing to comply with study requirements, including continuous glucose monitoring, self-monitoring of blood glucose, lifestyle management, and insulin-based glycemic management.
7. Agreement to use effective contraception during the study.
8. Willingness to provide written informed consent.

Exclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus or other specific types of diabetes.
2. Receipt within 3 months prior to screening of premixed insulin therapy and/or basal-bolus insulin therapy and/or basal insulin plus OAD therapy for ≥7 cumulative days; or receipt within 1 year prior to screening of intensive insulin therapy (insulin pump or multiple daily injections); or receipt within 3 months prior to screening of GLP-1 receptor agonists; or inability to tolerate protocol-specified doses.
3. Known hypersensitivity or intolerance to study medications.
4. Acute diabetic complications (including diabetic ketoacidosis, hyperosmolar hyperglycemic state, or lactic acidosis).
5. Severe microvascular complications: proliferative diabetic retinopathy; albumin excretion rate (AER) >300 mg/g or proteinuria >0.5 g/day; uncontrolled painful diabetic neuropathy or significant autonomic neuropathy. Severe macrovascular complications: hospitalization for acute cerebrovascular accident, acute coronary syndrome, peripheral artery disease requiring intervention or amputation within the previous 12 months; unstable angina, myocardial infarction, uncontrolled arrhythmia, or severe heart failure (New York Heart Association [NYHA] class ≥III).
6. Persistent blood pressure >180/110 mmHg, or uncontrolled above 160/110 mmHg within 1 week.
7. Estimated creatinine clearance <45 mL/min/1.73 m² (calculated by CKD-EPI formula); alanine aminotransferase ≥2.5 × upper limit of normal (ULN); or total bilirubin ≥1.5 × ULN.
8. Hemoglobin <100 g/L or requiring regular blood transfusions.
9. Use within 12 weeks prior to screening of medications affecting glycemic control for >1 cumulative week, including oral/intravenous glucocorticoids, growth hormone, estrogen/progestins, high-dose diuretics, or antipsychotics. Exceptions: low-dose diuretics used for antihypertensive purposes (HCTZ <25 mg/day, indapamide ≤1.5 mg/day) and physiological thyroid hormone replacement therapy.
10. Uncontrolled endocrine disorders.
11. History or family history of medullary thyroid carcinoma, or history of multiple endocrine neoplasia syndrome type 2 (MEN2).
12. Psychiatric illness or communication disorders.
13. Systemic infection, severe comorbid conditions, malignancy, or chronic diarrhea.
14. Pregnancy, lactation, or women of childbearing potential unwilling to use contraception during the study.
15. Uncooperative participants, inability to comply with follow-up, or judged by investigators as unlikely to complete the study.
16. Any other condition deemed unsuitable by investigators, including history of acute pancreatitis, rapidly progressing gallstones, or chronic cholecystitis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with optimal glycemic control | 24 weeks
  proportion of patients achieving glycosylated hemoglobin A1C <7% at 24 weeks in each treatment group.

SECONDARY OUTCOMES:
Proportion of subjects with excellent glycemic control | 24 weeks
  proportion of patients achieving glycosylated hemoglobin A1C <6.5% at 24 weeks in each treatment group.
Proportion of subjects with glycemic control | 48 weeks
  proportion of patients achieving glycosylated hemoglobin A1C <7% and <6.5% at 48 weeks in each treatment group.
Medication Compliance | 48 weeks
  differences in proportion of patients continuing the assigned regimen at 48 weeks in each treatment group.
Incidence of adverse events | 24 weeks and 48 weeks
  differences in incident of weight gain, hypoglycemic events among treatment groups at 24 weeks and extension follow-up period.